CLINICAL TRIAL: NCT05709353
Title: A Randomised, Controlled Trial of MDMA-assisted Prolonged Exposure Therapy for Comorbid Alcohol Use Disorder and Post-traumatic Stress Disorder
Brief Title: MDMA-assisted Prolonged Exposure Therapy for Comorbid Alcohol Use Disorder and Post-traumatic Stress Disorder
Acronym: MPATHY
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sydney (Other)
Collaborators: Monash University (Other); Sydney Local Health District (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: X22-0121
Record Dates: First submitted 2023-01-20; First posted 2023-02-02 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: PTSD; Alcohol Use Disorder; Alcohol Dependence; Post-traumatic Stress Disorder; Comorbidities and Coexisting Conditions
Keywords: MDMA-assisted therapy; Randomised-Controlled Trial; Comorbid PTSD and AUD; MDMA; COPE; Concurrent Treatment of PTSD and Substance Use Disorders Using Prolonged Exposure; Psychedelic-Assisted Therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Alcoholism | interventions — N-Methyl-3,4-methylenedioxyamphetamine; Niacin; Niacinamide

STUDY DESIGN:
Intervention Model Description: Randomised, double-blind between group comparison of change in PTSD symptoms and alcohol consumption
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COPE + MDMA (Experimental): 4x COPE sessions
  Dose 1:
  2x MDMA capsules (80mg) + 1x niacin-matched placebo capsule
  Optional supplementary dispense:
  1x MDMA capsule (40mg)
  4x COPE sessions
  Dose 2:
  2x MDMA capsules (80mg) + 1x niacin-matched placebo capsule
  Optional supplementary dispense:
  1x OR 2x white MDMA capsule (40 or 80mg)
  4x COPE sessions
  Interventions: Behavioral: Prolonged exposure therapy; Drug: MDMA
- COPE + Niacin (Control) (Other): 4x COPE sessions
  Dose 1:
  2x MDMA-matched placebo capsules + 1x niacin capsule (250mg)
  Optional supplementary dispense:
  1x MDMA-matched placebo capsule
  4x COPE sessions
  Dose 2:
  2x MDMA-matched placebo capsules + 1x niacin capsule (250mg)
  Optional supplementary dispense:
  1x OR 2x MDMA-matched placebo capsule
  4x COPE sessions
  Interventions: Behavioral: Prolonged exposure therapy; Drug: Niacin

INTERVENTIONS:
Behavioral: Prolonged exposure therapy — COPE represents an integration of existing evidence-based manualised CBT interventions for PTSD and substance dependence (see manual DOI: 10.1093/med:psych/9780199334513.001.0001). COPE used in the current study will represent an integration of existing evidence-based manualised CBT interventions for PTSD and substance dependence. COPE only begins when the participant in a safe environment and no longer in contact with the traumatic event/exposure.
  COPE employs imaginal and in vivo exposures to treat PTSD and consists of 12 individual 90-minute sessions (i.e. 19.5 hours) delivered by a clinical psychologist.
  Other Names: COPE (Concurrent Treatment of PTSD and Substance Use Disorders Using Prolonged Exposure)
Drug: MDMA — Administration of 80 to 160 mg MDMA across two 'dosing' sessions. Supplemental doses (additional 40mg during first session, additional 40- 80mg during second session) will be dependent on clinician and participant consensus during preparatory period of 'dosing session'. These supplemental amounts will be dispensed 60 to 90 minutes after initial 80 mg dose.
  Other Names: 3,4-Methyl enedioxy methamphetamine
  Arms: COPE + MDMA
Drug: Niacin — Administration of niacin 250mg or niacin-matched placebo during two 'dosing' sessions.
  Other Names: Control, Vitamin B3
  Arms: COPE + Niacin (Control)

SUMMARY:
To explore the effectiveness of of MDMA-assisted prolonged exposure therapy in improving treatment outcomes for individuals with comorbid PTSD and alcohol use disorder in a double-blind randomised placebo-controlled trial.

DETAILED DESCRIPTION:
New strategies for the treatment of comorbid PTSD and alcohol dependence are urgently required. Recent evidence has shown strong support for trauma-focused integrated treatments (namely COPE), however, only 49% demonstrate clinically significant improvements. MDMA may be a promising approach to improve response to COPE for this population. Emerging evidence suggests that MDMA-assisted therapy may be of promise for PTSD, and has demonstrated a good safety profile and potential efficacy in alcohol dependence.

This project will evaluate the clinical efficacy and tolerability of MDMA-assisted COPE relative to a control-assisted COPE. Active control used in this study is niacin. The investigators hypothesise that MDMA treated participants will be have a reduction in PTSD symptom severity as well as heavy drinking.

The trial will utilise a double blind, randomised, controlled design. A sample of 120 individuals will receive 14 weeks of treatment including 12 COPE sessions and 2 dosing sessions with MDMA (80-160mg) or control (niacin 250mg).

ELIGIBILITY:
Inclusion Criteria:

1. Both AUD and current PTSD according to the DSM-5 criteria, for 6 months or longer with at least moderate severity, according to investigator judgement and CAPS-5
2. Aged ≥18 years old
3. Adequate cognition and English language skills to give valid consent and complete research interviews assessments
4. Willing to give written informed consent
5. Received prior treatment for PTSD or AUD (not including study interventions)
6. Stable housing
7. Able to identify a significant other (such as a family/friend/partner) who could accompany them from clinic/provide transport and/or be contacted by the study team if required

Exclusion Criteria:

1. History of, or currently meeting, DSM-5 criteria for:

   * current or lifetime psychotic or bipolar disorders, or
   * major depression with psychotic features Assessed via Structured Clinical Interview for DSM-5 - Research Version (SCID-5-RV). Potential participants will be screened for personality disorders but suitability will then be confirmed by clinical interview given the prevalence of high scores in this comorbid population
2. Pregnant or lactating (contraception must be used and a sensitive pregnancy test will be performed at baseline and prior to dosing)
3. Significant alcohol withdrawal (current Clinical Institute Withdrawal Assessment for Alcohol [CIWA-Ar] score ≥10, including history of delirium tremens or alcohol withdrawal seizures).
4. Concurrent use of psychotropic medication (antidepressants and alcohol pharmacotherapy use considered if assessed by physician and titrated down with 5 half-lives + 1 week washout)
5. Use of, and unable or unwilling to cease, any medications likely to interact with MDMA in the opinion of the physicians and investigators during the trial (low dose opiates are permitted for pain management but not the night before or after MDMA sessions)
6. Substance use disorder other than tobacco (e.g. benzodiazepines, cannabis)
7. Abnormal clinical findings including a history of, or current: cardiac disease and/or dysrhythmia, uncontrolled hypertension or severe hypotension, abnormal electrocardiogram findings, stroke, liver disease, a history of epilepsy, hyponatraemia, or malignant hyperthermia (controlled hypertension and diabetes type II may be permitted)
8. Suicide risk according to clinician judgement and responses to Columbia Suicide Severity Rating Scale-Lifetime (C-SSRS-L) and SCID-5-RV.

   • Details surrounding any previous attempts >6 months ago will be gathered whereby attempts related to their trauma/PTSD and/or associated with the use of psychostimulants will contribute to risk assessment and guide trial safety measures if enrolled
9. Clinically unstable systemic medical (e.g., cancer) or psychiatric disorder or condition that might require hospitalisation that precludes trial participation
10. Regular use of ecstasy (e.g. at least twice in last 6 months, or >10 times within the last 5 years)
11. Enrolled in any other interventional clinical trials in the previous two months or over the duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-09-19 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
change in clinician-rated PTSD severity via Clinician-Administered PTSD Scale for DSM-5 (Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition) (CAPS-5) from baseline to visit 16. | 52 weeks
  CAPS-5 is a structured diagnostic interview with excellent psychometric properties and diagnostic efficiency and used widely in MDMA-assisted PTSD studies. The CAPS-5 will be administered by independent evaluators blind to treatment condition.
  CAPS-5 total symptom severity score is calculated by summing severity scores for the 20 DSM-5 PTSD symptoms.
  CAPS-5 symptom cluster severity scores are calculated by summing the individual item severity scores for symptoms corresponding to a given DSM-5 cluster: Criterion B (items 1-5); Criterion C (items 6-7); Criterion D (items 8-14); and, Criterion E (items 15-20).
change in self-reported PTSD symptom severity via Post-Traumatic Stress Disorder Checklist for DSM-5 (Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition) (PCL-5) from baseline to visit 16. | 52 weeks
  PCL-5 has excellent psychometric characteristics for a secondary indicator of PTSD symptom severity.
  Items are summed to provide a total severity score (range = 0-80). The PCL-5 can determine a provisional diagnosis in two ways: Summing all 20 items (range 0-80) and using a cut-point score of 31-33 appears to be reasonable based upon current psychometric work.

SECONDARY OUTCOMES:
Number of Heavy Drinking Days per week (HDDs) (>5 standard drinks/day for men; >4 for women) | 52 weeks
  This will be measured by the Timeline Follow Back and corroborated with Phosphatidylethanol (PEth) levels
Absence of any HDD | 52 weeks
  Measured by Timeline Follow Back and corroborated with Phosphatidylethanol (PEth) levels

OTHER OUTCOMES:
Mean alcohol consumption per drinking day | 52 weeks
  Measured by Timeline Follow Back and corroborated with Phosphatidylethanol (PEth) levels
Change in dependence Severity | 52 weeks
  Measured by the Alcohol Dependence Scale. The minimum score is 0 and the maximum score is 47. A higher score indicates more severe dependence.
Changes in Anxiety | 52 weeks
  Measured by cumulative scores on the DASS-21 Anxiety Scale. This scale has a minimum score of 0 and maximum score of 21. A higher score indicates more anxiety.
Changes in Depression | 52 weeks
  Measured by cumulative scores on the DASS-21 Depression Scale. This scale has a minimum score of 0 and maximum score of 21. A higher score indicates greater depression.
Changes in Stress | 52 weeks
  Measured by cumulative scores on the DASS-21 Stress Scale. This scale has a minimum score of 0 and maximum score of 21. A higher score indicates more stress.
Sleep Disturbances | 52 weeks
  As measured by the ISI (Insomnia Severity Index). This Index has a minimum score of 0 and a maximum score of 28. The higher the score indicates more severe insomnia.
Drinking Diary | 16 weeks
  Daily texts will be sent out to participants querying the amount of alcohol they have consumed. Participant responses to this will be recorded. This will be managed through SEMA software.
Mood states | 16 weeks
  Daily texts will be sent out to participants querying their moods. This will be in line with the POMS instrument (Profile of Mood States).
Mood following dosing session | week 5, week 10
  The week following each dosing session will involve calls with participants to complete POMS (profile of mood states)
Changes in Suicidal Ideation | 52 weeks
  Changes in suicidal ideation & behaviours across the treatment period. This will be measured on the C-SRSS (Columbia Suicide Severity Rating Scale). At baseline this will be measured by the baseline version. At each visit following this, this will be recorded on the since last visit version. Higher scores indicate more severe suicidality.
Changes in Quality of Life | 16 weeks
  To assess whether treatment can change quality of life as measured by the short form Health Survey (SF-36). This survey has 36 items that measure 8 domains of health, including: physical functioning, physical role limitations, bodily pain, general health perceptions, energy/vitality, social functioning, emotional role limitations and mental health. The scores are transformed to range from 0 (worst possible health) to 100 (best possible health).
Changes PTSD cognitions | 52 weeks
  As measured by the PTCI. This is a 33 question inventory measures negative cognitions about the self & world, as well as self-blame. Higher scores indicate more negative cognitions.
Changes in use of Health Services | 16 weeks
  As measured by the Brief Health Services Use Questionnaire. This questionnaire assesses Health Service Use across the last 3 months. It is a qualitative questionnaire.
Therapeutic Alliance between therapist | 16 weeks
  As measured by the Helping Alliance Questionnaire (HAQ-II). This instrument will be completed by the patient (patient version) and the clinician (clinician version). This outlines how a person may feel or behave in relation to their therapist. Higher scores indicates a better therapeutic alliance.
COPE Session Rating Scale | 16 weeks
  As measured by the session rating scale (SRS). Following each COPE session, both the therapist and participant will complete a brief post-session rating. This scale measures; relationship, goals & topics, approach or method and overall psychotherapy session. Higher scores on each of these indicate a more positive experience.
Treatment Satisfaction as measured by the YES (your experience of service). | 16 weeks
  This instrument is designed to gather information from consumers about their experiences of care.
Treatment Satisfaction ss measured by the CSQ-8 (client satisfaction questionnaire). | 16 weeks
  This instrument measures clients satisfaction with treatment. Total scores range from 8 to 32, with the higher number indicating greater satisfaction.
Measurement of Distress ss measured by a Likert Scale | week 5, week 12
  This instrument will be administered hourly within the dosing sessions. It aims to measure the participant's mood on a scale of 1 (worst) -10 (best)
Measurement of Drug Effect as measured by the Revised Mystical Experience Questionnaire 30 (MEQ-30) | week 5, week 12
  MEQ-30 Measures mystical, positive mood, transcendence, ineffability experienced in dosing sessions.
  MEQ-30 will be compelted at the end of each dosing session. participants will be asked to rate rate the degree to which at any time during that session they experienced certain phenomena on a scale of 0 (not at all) to 5 (more than any other time in their life)

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten C Morley, PhD, Principal Investigator — University of Sydney
Locations (2):
- Australia (2):
  - Drug Health Services, Royal Prince Alfred Hospital, Sydney, New South Wales
  - Turning Point, Richmond, Victoria

IPD SHARING:
Plan to Share IPD: No